CLINICAL TRIAL: NCT01463098
Title: A 2-Part, Randomized, Double-Blind, Placebo- and Active- Controlled, Single Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2006 in Healthy Subjects and Otherwise Healthy Subjects With Primary Insomnia
Brief Title: A 2-Part Single Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2006-A001-001
Record Dates: First submitted 2011-10-26; First posted 2011-11-01 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2013-03

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — lemborexant; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (14):
- Part A: E2006 1.0 mg (Experimental)
  Interventions: Drug: E2006 1.0 mg
- Part A: E2006 2.5 mg (Experimental)
  Interventions: Drug: E2006 2.5 mg
- Part A: E2006 5.0 mg (Experimental)
  Interventions: Drug: E2006 5.0 mg
- Part A: E2006 10.0 mg (Experimental)
  Interventions: Drug: E2006 10.0 mg
- Part A: E2006 25.0 mg (Experimental)
  Interventions: Drug: E2006 25.0 mg
- Part A: E2006 50.0 mg (Experimental)
  Interventions: Drug: E2006 50.0 mg
- Part A: E2006 100 mg (Experimental)
  Interventions: Drug: E2006 100 mg
- Part A: E2006 200 mg (Experimental)
  Interventions: Drug: E2006 200 mg
- Part B: Zolpidem 10 mg (Experimental)
  Interventions: Drug: Zolpidem 10 mg
- Part B: E2006 Matched Placebo or Zolpidem Matched Placebo (Experimental)
  Interventions: Drug: E2006 Matched Placebo or Zolpidem Matched Placebo
- Part A: E2006 Matched Placebo (Experimental)
  Interventions: Drug: E2006 Matched Placebo
- Part B: E2006 2.5 mg (Experimental)
  Interventions: Drug: E2006 2.5 mg
- Part B: E2006 10 mg (Experimental)
  Interventions: Drug: E2006 10.0 mg
- Part B: E2006 25 mg (Experimental)
  Interventions: Drug: E2006 25.0 mg

INTERVENTIONS:
Drug: E2006 1.0 mg — E2006 1.0 mg capsule.
  Other Names: Lemborexant
  Arms: Part A: E2006 1.0 mg
Drug: E2006 2.5 mg — E2006 2.5 mg capsule.
  Other Names: Lemborexant
  Arms: Part A: E2006 2.5 mg; Part B: E2006 2.5 mg
Drug: E2006 5.0 mg — E2006 5.0 mg (2 capsules of 2.5 mg each).
  Other Names: Lemborexant
  Arms: Part A: E2006 5.0 mg
Drug: E2006 10.0 mg — E2006 10.0 mg capsule.
  Other Names: Lemborexant
  Arms: Part A: E2006 10.0 mg; Part B: E2006 10 mg
Drug: E2006 25.0 mg — E2006 25.0 mg (2 capsules of 10 mg each and 2 capsules of 2.5 mg each).
  Other Names: Lemborexant
  Arms: Part A: E2006 25.0 mg; Part B: E2006 25 mg
Drug: E2006 50.0 mg — E2006 50.0 mg capsule.
  Other Names: Lemborexant
  Arms: Part A: E2006 50.0 mg
Drug: E2006 100 mg — E2006 100 mg (2 capsules of 50 mg each).
  Other Names: Lemborexant
  Arms: Part A: E2006 100 mg
Drug: E2006 200 mg — E2006 200 mg (4 capsules of 50 mg each).
  Other Names: Lemborexant
  Arms: Part A: E2006 200 mg
Drug: Zolpidem 10 mg — Zolpidem 10 mg immediate release tablet.
  Arms: Part B: Zolpidem 10 mg
Drug: E2006 Matched Placebo or Zolpidem Matched Placebo — E2006-matched placebo capsules or zolpidem-matched placebo tablets.
  Arms: Part B: E2006 Matched Placebo or Zolpidem Matched Placebo
Drug: E2006 Matched Placebo — E2006-matched placebo capsule.
  Arms: Part A: E2006 Matched Placebo

SUMMARY:
Part A: The purpose of this study is to evaluate the safety and tolerability of single oral doses of E2006 administered in the morning to healthy male and female subjects.

Part B: The purpose of this study is to evaluate selected pharmacodynamic (PD) parameters (e.g., polysomnographically defined sleep measures) with regard to dose response in subjects with primary insomnia following single oral dosing of E2006 in the evening approximately 30 minutes prior to the sleep period, compared with 10 mg zolpidem and placebo.

ELIGIBILITY:
Key Inclusion Criteria:

Healthy Subjects:

* With habitual time in bed > 7 hours, with lights out 2200 to 2400 and lights on 0600 to 0800
* Who report typical sleep latency of </= 30 minutes
* With typical total sleep time (TST) >/= 420 minutes

Primary Insomnia Subjects:

* Otherwise healthy adult male and female subjects with a diagnosis of primary insomnia (as defined by the Diagnostic and Statistical Manual of Mental Disorders-IV-Text Revision [DSM-IV-TR]) present at the time of Screening for at least 3 months
* With a score of > 15 on the Insomnia Severity Index (ISI) at Screening
* Who report taking >/= 30 minutes to fall asleep on at least 3 nights per week for the past month
* Who report 6.5 hours sleep or less on at least 3 nights per week for the past month
* With mean latency to persistent sleep (LPS) on both baseline nights of >/= 20 minutes with neither night < 15 minutes
* With mean wake after sleep onset (WASO) >/= 20 minutes on both baseline nights, with neither night < 15 minutes or mean TST > 420 minutes

Key Exclusion Criteria:

* With a current history of sleep disorders (e.g., obstructive sleep apnea, restless leg syndrome [RLS], narcolepsy, or circadian rhythm disorder) other than primary insomnia (for Part B)
* Subjects with any clinically abnormal symptom or organ impairment found in medical history, symptoms/signs, vital signs, ECG finding, or laboratory test results which require medical treatment
* All females must be of non-childbearing potential
* With a known history of significant neurological or serious psychiatric illness

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2011-10-05 (Actual); Primary Completion 2012-08-11 (Actual); Study Completion 2012-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinilabs, Inc., New York, New York
  - Community Research, Cincinnati, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in United States from 05 October 2011 to 11 August 2012.
Pre-assignment Details: Part A: A total of 160 healthy participants were screened, of which 96 were screen failures and 64 were enrolled and randomized to receive study treatment.
  Part B: A total of 281 otherwise healthy participants with primary insomnia were screened, of which 223 were screen failures and 58 were enrolled and randomized to receive study treatment.
Groups:
- Part A: E2006 Matched Placebo: Healthy participants received E2006-matched placebo, capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 1.0 mg: Healthy participants received E2006 1 milligram (mg), capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 2.5 mg: Healthy participants received E2006 2.5 mg, capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 5 mg: Healthy participants received E2006 5 mg (2 capsules of 2.5 mg each), orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 10 mg: Healthy participants received E2006 10 mg, capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 25 mg: Healthy participants received E2006 25 mg (2 capsules of 10 mg each and 2 capsules of 2.5 mg each), orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 50 mg: Healthy participants received E2006 50 mg, capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 100 mg: Healthy participants received E2006 100 mg (2 capsules of 50 mg each), orally in the morning, one hour after lights-on, on Day 1.
- Part A: E2006 200 mg: Healthy participants received E2006 200 mg (4 capsules of 50 mg each), orally in the morning, one hour after lights-on, on Day 1.
- Part B: E2006 Matched Placebo or Zolpidem Matched Placebo: Otherwise healthy participants with primary insomnia received E2006-matched placebo capsules or zolpidem-matched placebo tablets, orally in the evening, 30 minutes prior to habitual bed time (lights-out) on Day 1.
- Part B: Zolpidem 10 mg: Otherwise healthy participants with primary insomnia received zolpidem 10 mg immediate release, tablet, orally in the evening, 30 minutes prior to habitual bed time (lights-out) on Day 1.
- Part B: E2006 2.5 mg: Otherwise healthy participants with primary insomnia received E2006 2.5 mg, capsule, orally in the evening, 30 minutes prior to habitual bed time (lights-out) on Day 1.
- Part B: E2006 10 mg: Otherwise healthy participants with primary insomnia received E2006 10 mg, capsule, orally in the evening, 30 minutes prior to habitual bed time (lights-out) on Day 1.
- Part B: E2006 25 mg: Otherwise healthy participants with primary insomnia received E2006 25 mg (2 capsules of 10 mg each and 2 capsules of 2.5 mg each), orally in the evening, 30 minutes prior to habitual bed time (lights-out) on Day 1.
Period: Part A (11 Days)
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 14 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 5 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Choice | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (11 Days)
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11 | 13 | 10 | 12
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 11 | 12 | 10 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant Choice | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received study drug and had at least one post dose safety assessment.
Groups:
- Part A: E2006 1.0 mg: Healthy participants received E2006 1 mg, capsule, orally in the morning, one hour after lights-on, on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 11 | 13 | 10 | 12 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 11 | 13 | 10 | 12 | 122
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 4 | 6 | 59
  Male | 8 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 7 | 6 | 6 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 2 | 1 | 1 | 2 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 18
  Not Hispanic or Latino | 14 | 4 | 5 | 4 | 5 | 5 | 4 | 3 | 3 | 12 | 11 | 12 | 10 | 12 | 104
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 6 | 3 | 2 | 3 | 2 | 4 | 2 | 2 | 2 | 6 | 2 | 7 | 4 | 5 | 50
  White | 8 | 3 | 3 | 3 | 2 | 2 | 2 | 3 | 4 | 6 | 8 | 6 | 5 | 7 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Treatment Emergent Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs)
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  AEs | 7 | 1 | 0 | 1 | 4 | 2 | 4 | 2 | 5
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part A: Number of Participants With Markedly Abnormal Laboratory Parameter Values
Time Frame: Baseline up to Day 6
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 6 | 1 | 3 | 1 | 2 | 2 | 3 | 1 | 0

3. Primary Outcome: Part A: Number of Participants With Significant Change From Baseline in Vital Sign Values
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Parameter Values
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part A: Number of Participants With Any Suicidality Assessed Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess any suicidality, any suicidal behavior, any suicidal ideation. Any suicidality: emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior: when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: when response is "yes" for any of these questions- wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide. Number of Participants with any suicidality has been reported for this outcome measure.
Time Frame: Baseline, Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B: Change From Baseline in Latency to Persistent Sleep (LPS) Assessed Using Polysomnography (PSG) Measurement at Day 1
Description: LPS was the duration of time in minutes from lights off to the first 30 seconds of recording (epoch) of 20 consecutive epochs of non-wakefulness as measured by PSG.
Time Frame: Baseline, Day 1
Population: Pharmacodynamic (PD) analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Baseline | 56.3 (20.5) | 51.8 (26.7) | 50.1 (35.1) | 55.9 (40.5) | 62.8 (38.3)
  Change From Baseline at Day 1 | -7.17 (30.9) | -33.1 (20.3) | -28.1 (45.2) | -28.8 (39.0) | -43.9 (35.9)

7. Primary Outcome: Part B: Change From Baseline in Total Sleep Time (TST) Assessed Using PSG at Day 1
Description: TST was the duration in minutes including rapid eye movement (REM) sleep plus non-rapid eye movement (NREM) sleep during the time spent in bed.
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Baseline | 335 (56.2) | 349 (49.9) | 341 (46.7) | 345 (60.7) | 342 (46.9)
  Change From Baseline at Day 1 | 14.0 (47.6) | 61.3 (41.9) | 51.9 (60.5) | 61.8 (34.0) | 85.8 (49.9)

8. Primary Outcome: Part B: Change From Baseline in Sleep Efficiency Assessed Using PSG at Day 1
Description: Sleep efficiency was defined as the TST divided by the time in bed (minutes) multiplied by 100. TST was the duration in minutes including REM sleep plus NREM sleep during the time spent in bed.
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: percentage of time asleep
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
percentage of time asleep
  Baseline | 69.8 (11.7) | 72.7 (10.4) | 71.1 (9.72) | 71.9 (12.6) | 71.3 (9.77)
  Change From Baseline at Day 1 | 2.90 (9.93) | 12.8 (8.73) | 10.8 (12.6) | 12.9 (7.08) | 17.9 (10.4)

9. Primary Outcome: Part B: Change From Baseline in Wake After Sleep Onset (WASO) Assessed Using PSG at Day 1
Description: WASO was defined as the duration (in minutes) of wakefulness from onset of persistent sleep to lights-on.
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Baseline | 95.7 (52.9) | 85.7 (39.6) | 95.6 (41.5) | 84.7 (64.0) | 85.4 (20.7)
  Change From Baseline at Day 1 | -7.52 (27.3) | -32.1 (30.7) | -28.9 (59.0) | -28.3 (53.6) | -45.6 (21.1)

10. Primary Outcome: Part B: Change From Baseline in Number of Awakenings After Persistent Sleep (NAW) Assessed Using PSG at Day 1
Description: Number of awakenings was determined from LPS to lights-on. LPS was the duration of time measured from lights off to the first 30 seconds of PSG measurement recording (epoch) of 20 consecutive epochs of non-wake. An awakening was defined as a PSG recording of at least two consecutive wake epochs.
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: awakenings
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
awakenings
  Baseline | 10.5 (3.91) | 12.4 (5.33) | 11.9 (3.48) | 12.3 (4.08) | 10.9 (3.52)
  Change From Baseline at Day 1 | 0.125 (3.48) | -3.45 (3.08) | -1.38 (4.87) | -0.30 (6.85) | 0.542 (4.17)

11. Primary Outcome: Part B: Change From Baseline in Percentage of Each Sleep Stage Duration Assessed Using PSG at Day 1
Description: Sleep stages included NREM sleep and REM (dreaming) sleep. Non-REM sleep is comprised of the sum of Stage N1 (light sleep), N2 (also fairly light, with sudden increases in brain wave frequency known as sleep spindles) and N3 or slow wave sleep (deep sleep). Sleep was staged in sequential 30-second epochs.
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: percentage of sleep stage duration
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
percentage of sleep stage duration
  Stage N1: Baseline | 11.8 (5.74) | 10.3 (3.47) | 15.2 (5.70) | 11.9 (4.44) | 11.5 (2.54)
  Stage N1: Change at Day 1 | 0.00429 (5.29) | -0.715 (5.02) | -4.28 (6.11) | 2.19 (4.92) | -2.67 (2.49)
  Stage N2: Baseline | 56.5 (7.73) | 56.3 (6.70) | 57.5 (10.9) | 60.6 (12.0) | 51.5 (6.61)
  Stage N2: Change at Day 1 | 0.390 (4.64) | -0.316 (4.96) | -0.306 (7.49) | -3.12 (9.36) | -2.73 (5.77)
  Stage N3/Slow Wave Sleep: Baseline | 14.0 (8.74) | 15.0 (9.77) | 10.9 (9.78) | 11.8 (12.1) | 17.2 (4.75)
  Stage N3/Slow Wave Sleep : Change at Day 1 | 0.0613 (2.90) | 2.15 (3.77) | -0.0852 (6.10) | 1.01 (8.55) | -0.42 (3.28)
  Stage REM: Baseline | 17.7 (4.86) | 18.4 (4.59) | 16.4 (3.52) | 15.7 (3.46) | 19.8 (4.93)
  Stage REM: Change at Day 1 | -0.455 (3.58) | -1.12 (4.13) | 4.67 (6.54) | -0.0712 (7.07) | 5.82 (5.27)

12. Primary Outcome: Part B: Change From Baseline in Duration (in Minutes) of Each Sleep Stage Assessed Using PSG at Day 1
Description: as for outcome 11
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Stage N1: Baseline | 37.8 (16.6) | 35.1 (11.3) | 50.1 (15.5) | 40.7 (17.3) | 38.9 (11.0)
  Stage N1: Change at Day 1 | 2.38 (17.8) | 3.41 (17.4) | -7.65 (15.0) | 14.7 (19.9) | -1.35 (11.1)
  Stage N2: Baseline | 190 (39.4) | 195 (27.7) | 198 (52.7) | 212 (63.6) | 175 (29.2)
  Stage N2: Change at Day 1 | 10.4 (34.3) | 34.4 (33.9) | 29.6 (52.3) | 21.5 (38.8) | 33.6 (36.6)
  Stage N3/Slow Wave Sleep: Baseline | 47.7 (33.2) | 53.4 (35.2) | 36.5 (32.1) | 38.3 (37.8) | 59.1 (18.2)
  Stage N3/Slow Wave Sleep: Change at Day 1 | 1.94 (12.7) | 16.3 (17.4) | 3.73 (18.3) | 14.9 (28.8) | 12.7 (11.3)
  Stage REM: Baseline | 59.4 (19.3) | 65.3 (20.0) | 56.7 (15.7) | 54.0 (14.0) | 68.8 (19.6)
  Stage REM: Change at Day 1 | -0.729 (13.3) | 7.14 (19.2) | 26.3 (31.8) | 10.7 (29.5) | 40.8 (21.7)

13. Primary Outcome: Part B: Change From Baseline in Mean Total Number of Shift in Sleep Stages Assessed Using PSG at Day 1
Description: as for outcome 11
Time Frame: Baseline, Day 1
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: stage shift
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
stage shift
  Baseline | 167 (22.3) | 168 (35.5) | 174 (42.2) | 188 (45.6) | 153 (36.7)
  Change From Baseline at Day 1 | 0.250 (35.7) | 4.18 (41.2) | -16.3 (30.4) | 14.4 (53.1) | 14.0 (28.1)

14. Primary Outcome: Part B: Change From Day 1 in Waketime Questionnaire Parameters: How Long Did You Sleep Last Night at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm anticipated reports of poor sleep. In this outcome measure, data for question "How long did you sleep last night" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Day 1 | 302.1 (82.39) | 292.3 (61.21) | 298.8 (106.45) | 302.5 (71.70) | 276.3 (82.77)
  Change From Day 1 at Day 6 | -3.3 (74.66) | 12.7 (55.11) | 42.4 (89.08) | -41.5 (87.24) | 20.0 (60.11)

15. Primary Outcome: Part B: Change From Day 1 in Waketime Questionnaire Parameters: Time to Fall Asleep Last Night at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm anticipated reports of poor sleep. In this outcome measure, data for question "Time to fall asleep last night" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Day 1 | 70.8 (22.55) | 67.3 (30.36) | 72.2 (51.99) | 82.5 (61.02) | 108.1 (65.00)
  Change From Day 1 at Day 6 | 8.3 (36.33) | 9.1 (28.09) | -3.8 (31.37) | 46.5 (76.63) | -13.7 (42.57)

16. Primary Outcome: Part B: Change From Day 1 in Waketime Questionnaire Parameters: Number of Awakening After Falling Asleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm anticipated reports of poor sleep. In this outcome measure, data for question "Number of awakening after falling asleep" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
number of awakenings
  Day 1 | 2.7 (1.30) | 2.7 (1.42) | 2.8 (1.30) | 2.7 (1.42) | 3.6 (1.24)
  Change From Day 1 at Day 6 | -0.1 (1.16) | -0.3 (1.10) | -0.6 (1.39) | 0.7 (2.31) | 0.3 (0.97)

17. Primary Outcome: Part B: Change From Day 1 in Waketime Questionnaire Parameters: Time Spent Awake After Falling Asleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm anticipated reports of poor sleep. In this outcome measure, data for question "Time spent awake after falling asleep" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
minutes
  Day 1 | 133.8 (115.76) | 101.8 (76.36) | 82.3 (46.31) | 102.0 (68.56) | 128.8 (88.30)
  Change From Day 1 at Day 6 | -27.9 (136.39) | -5.5 (55.70) | -3.7 (54.03) | 46.8 (140.47) | 10.7 (93.91)

18. Primary Outcome: Part B: Change From Day 1 in Waketime Questionnaire Parameters: Rate Quality of Your Sleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm anticipated reports of poor sleep. In this outcome measure, data for question "Rate quality of your sleep" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
score on a scale
  Day 1 | 2.8 (0.72) | 3.1 (0.83) | 2.6 (0.65) | 2.6 (0.70) | 2.8 (0.75)
  Change From Day 1 at Day 6 | -0.6 (0.67) | -0.5 (0.93) | -0.5 (0.78) | 0.2 (0.92) | -0.4 (1.00)

19. Primary Outcome: Part B: Change From Day 1 (Pre-dose) in Digit Symbol Substitution Test (DSST) Score at Day 6
Description: DSST is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the participant to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than cognitive functioning) to 133 (greater than cognitive functioning) as a description of DSST. An increase in score represents an improvement in an integrated measure of cognitive function.
Time Frame: Day 1 (Pre-dose), Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
score on a scale
  Day 1 (Pre-dose) | 53.0 (9.56) | 50.7 (11.64) | 48.2 (10.80) | 51.0 (6.48) | 49.5 (11.87)
  Change From Day 1 (Pre-dose) at Day 6 | 9.8 (15.15) | 10.5 (14.44) | 14.3 (13.34) | 8.3 (15.33) | 11.7 (20.67)

20. Primary Outcome: Part B: Change From Day 1 (Pre-dose) in Number of Lapses of Greater Than (>) 500- Milliseconds (Msec) Assessed by Psychomotor Vigilance Test (PVT) at Day 6
Description: PVT, a computer-based test, is a chronometric measure of an individual's reaction to specified small changes in a labile environment. Participants were instructed to respond to a digital signal on a computer terminal by pressing a key. Errors of omission and commission are recorded. When a participant did not respond to the PVT signal within 500 msec, it was termed a lapse. The higher the number of lapses the greater the impairment.
Time Frame: Day 1 (Pre-dose), Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: lapses
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
lapses
  Day 1 (Pre-dose): number analyzed (Participants) | 12 | 11 | 12 | 10 | 12
  Day 1 (Pre-dose) | 2.3 (3.67) | 3.0 (2.86) | 4.1 (7.57) | 4.4 (4.22) | 5.2 (12.00)
  Change From Day 1 (Pre-dose) at Day 6: number analyzed (Participants) | 12 | 11 | 12 | 10 | 12
  Change From Day 1 (Pre-dose) at Day 6 | 0.3 (2.49) | 2.3 (6.84) | 0.9 (5.33) | -1.4 (3.66) | -1.2 (9.57)

21. Primary Outcome: Part B: Change From Day 1 (Pre-dose) in Score on Karolinska Sleepiness Scale (KSS) at Day 6
Description: KSS is a 9-point scale, on which the participant has to mark his or her sleepiness during the previous 10 minutes. The scale ranges from 1, which indicates "extremely alert", to 9, which indicates "extremely sleepy, can't stay awake". Higher numbers indicating sleepier and lower numbers more alert.
Time Frame: Day 1 (Pre-dose), Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
score on a scale
  Day 1 (Pre-dose) | 4.4 (1.83) | 3.8 (2.04) | 4.0 (2.20) | 4.8 (2.20) | 5.5 (1.93)
  Change From Day 1 (Pre-dose) at Day 6 | -0.4 (1.68) | 1.0 (1.41) | 0.2 (1.34) | 0.3 (1.95) | -0.7 (2.27)

22. Secondary Outcome: Part A: Maximum Plasma Concentration (Cmax) of E2006
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: Pharmacokinetic (PK) analysis set included all participants who had sufficient PK data to derive at least one PK parameter. PK parameters for Part B were not analyzed due to change in planned analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 5.15 (27.1) | 14.9 (43.0) | 22.3 (19.1) | 32.0 (57.3) | 107 (20.3) | 161 (32.9) | 242 (47.0) | 429 (12.2)

23. Secondary Outcome: Part A: Time to Reach Maximum Plasma Concentration (Tmax) of E2006
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: PK analysis set included all participants who had sufficient PK data to derive at least one PK parameter. PK parameters for Part B were not analyzed due to change in planned analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.000 [1.00 to 1.08] | 1.010 [1.00 to 3.00] | 1.550 [0.92 to 3.00] | 1.000 [0.57 to 2.00] | 2.010 [1.00 to 3.00] | 2.525 [1.00 to 3.08] | 3.000 [3.00 to 5.00] | 3.000 [1.00 to 9.00]

24. Secondary Outcome: Part A: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC0-24) of E2006
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: PK analysis set included all participants who had sufficient PK data to derive at least one PK parameter. PK parameter for Part B were not analyzed due to change in planned analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
nanogram hour per milliliter (ng*h/mL) | 17.0 (17.5) | 53.8 (36.4) | 93.2 (18.9) | 150 (38.9) | 648 (15.4) | 1060 (33.0) | 1850 (33.8) | 3970 (24.8)

25. Secondary Outcome: Part A: Area Under the Plasma Concentration-time Curve From Time Zero to t Hours (AUC0-t) of E2006
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 18.4 (29.9) | 74.4 (45.9) | 126 (18.7) | 274 (30.4) | 1390 (31.3) | 1960 (38.5) | 4300 (35.1) | 9290 (39.5)

26. Secondary Outcome: Part A: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of E2006
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: PK analysis set included all participants who had sufficient PK data to derive at least one PK parameter. PK parameters for Part B were not analyzed due to change in planned analysis. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 5 | 4 | 5 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 19.5 (19.8) | 72.3 (54.3) | 146 (20.9) | 299 (31.7) | 1470 (33.7) | 2020 (40.3) | 4520 (36.8) | 9910 (39.5)

27. Secondary Outcome: Part A: Terminal Half-life (t1/2) of E2006 in Plasma
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
hours | 12.700 [9.12 to 65.10] | 30.100 [14.50 to 50.70] | 31.350 [26.20 to 42.80] | 56.150 [34.90 to 72.20] | 65.500 [53.60 to 71.60] | 51.850 [36.10 to 72.80] | 59.750 [50.50 to 73.00] | 65.200 [27.00 to 75.80]

28. Secondary Outcome: Part A: Apparent Total Clearance of E2006 From Plasma (CL/F)
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liter per hour (L/h) | 44.8 (39.0) | 28.2 (54.2) | 33.9 (18.6) | 33.4 (31.8) | 17.0 (33.4) | 24.8 (40.3) | 22.1 (36.9) | 20.2 (39.4)

29. Secondary Outcome: Part A: Apparent Volume of Distribution of E2006 in Plasma (Vz/F)
Time Frame: Day 1: Pre-dose, up to 240 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
liter (L) | 1170 (40.7) | 1200 (34.4) | 1610 (25.3) | 2670 (26.6) | 1580 (24.5) | 1810 (28.7) | 1930 (28.1) | 1680 (35.4)

30. Secondary Outcome: Part A: Cumulative Amount of Unchanged Drug E2006 Excreted Into the Urine (Ae)
Time Frame: Day 1: Pre-dose, up to 120 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram (mg)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
milligram (mg) | 0.000108 (28.6) | 0.0000777 (126) | 0.000667 (153) | 0.00141 (47.4) | 0.00788 (72.1) | 0.0113 (23.1) | 0.0307 (65.5) | 0.0402 (56.8)

31. Secondary Outcome: Part A: Renal Clearance (CLR) of Drug E2006
Time Frame: Day 1: Pre-dose, up to 120 hours post-dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute (mL/min)
Arm/Group | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
milliliter per minute (mL/min) | 0.0877 (29.8) | 0.0157 (70.7) | 0.0881 (129) | 0.0938 (68.7) | 0.111 (66.2) | 0.107 (34.5) | 0.140 (44.6) | 0.0844 (41.7)

32. Secondary Outcome: Part A: Maximum Change From Day 1 (Pre-dose) in Digit Symbol Substitution Test (DSST) Score at Day 6
Description: DSST is a cognitive test designed to assess psychomotor speed of performance requiring visual perception, spatial decision-making, and motor skills. It consists of 133 digits and requires the participant to substitute each digit with a simple symbol in a 90-second period. Each correct symbol is counted, and the total score ranges from 0 (less than cognitive functioning) to 133 (greater than cognitive functioning) as a description of DSST. An increase in score represents an improvement in an integrated measure of cognitive function. In this outcome measure, data for participants who received placebo matched to "1 mg, 2.5 mg, 5 mg E2006" and matched to "10 mg, 25 mg, 50 mg, 100 mg, and 200 mg E2006", has been presented separately.
Time Frame: Day 1 (Pre-dose), up to Day 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part A: Placebo: Matched to 1, 2.5, 5 mg E2006: Healthy participants received E2006-matched placebo (matched to 1 mg, 2.5 mg and 5 mg E2006), capsule, orally in the morning, one hour after lights-on, on Day 1.
- Part A: Placebo: Matched to 10, 25, 50, 100, 200 mg E2006: Healthy participants received E2006-matched placebo (matched to 10 mg, 25 mg, 50 mg, 100 mg, and 200 mg E2006), capsule, orally in the morning, one hour after lights-on, on Day 1.
Arm/Group | Part A: Placebo: Matched to 1, 2.5, 5 mg E2006 | Part A: Placebo: Matched to 10, 25, 50, 100, 200 mg E2006 | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
score on a scale
  Day 1 (Pre-dose) | 53.7 (13.84) | 59.1 (15.27) | 52.3 (10.33) | 63.7 (8.57) | 61.2 (13.53) | 60.5 (9.97) | 59.2 (8.06) | 59.8 (8.80) | 56.5 (8.57) | 62.8 (18.93)
  Maximum Change From Day 1 (Pre-dose) at Day 6: number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 4 | 6 | 5 | 6 | 6
  Maximum Change From Day 1 (Pre-dose) at Day 6 | 14.3 (14.01) | 7.8 (18.23) | 16.0 (11.42) | 9.0 (18.57) | 8.8 (18.81) | -9.0 (34.71) | 5.8 (30.01) | 2.6 (27.57) | -13.0 (18.97) | -16.3 (34.62)

33. Secondary Outcome: Part A: Maximum Change From Day 1 (Pre-dose) in Number of Lapses of > 500 Msec Assessed by Psychomotor Vigilance Test (PVT) at Day 6
Description: PVT, a computer-based test, is a chronometric measure of an individual's reaction to specified small changes in a labile environment. Participants were instructed to respond to a digital signal on a computer terminal by pressing a key. Errors of omission and commission are recorded. When a participant did not respond to the PVT signal within 500 msec, it was termed a lapse. The higher the number of lapses the greater the impairment. In this outcome measure, data for participants who received placebo matched to "1 mg, 2.5 mg, 5 mg E2006" and matched to "10 mg, 25 mg, 50 mg, 100 mg, and 200 mg E2006", has been presented separately.
Time Frame: Day 1 (Pre-dose), Day 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: lapses
Groups:
- Part A: Placebo: Matched to 1, 2.5, 5 mg E2006: Healthy participants received E2006-matched placebo (matched to 1 mg, 2,5 mg and 5 mg E2006), capsule, orally in the morning, one hour after lights-on, on Day 1.
Arm/Group | Part A: Placebo: Matched to 1, 2.5, 5 mg E2006 | Part A: Placebo: Matched to 10, 25, 50, 100, 200 mg E2006 | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
lapses
  Day 1 (Pre-dose) | 1.0 (0.89) | 1.8 (2.39) | 1.3 (2.42) | 2.5 (2.43) | 1.3 (1.97) | 1.5 (1.38) | 0.3 (0.52) | 2.5 (2.07) | 2.0 (1.90) | 6.5 (4.18)
  Maximum Change From Day 1 (Pre-dose) at Day 6: number analyzed (Participants) | 6 | 10 | 5 | 5 | 6 | 5 | 6 | 5 | 6 | 6
  Maximum Change From Day 1 (Pre-dose) at Day 6 | 6.0 (10.70) | 4.7 (3.37) | 3.4 (2.07) | 1.4 (4.45) | 2.5 (9.33) | 22.6 (10.45) | 19.7 (19.50) | 26.6 (12.42) | 29.2 (14.13) | 32.0 (16.63)

34. Secondary Outcome: Part A: Maximum Change From Day 1 (Pre-dose) in Karolinska Sleepiness Scale (KSS) Score at Day 6
Description: KSS is a 9-point scale, on which the participant has to mark his or her sleepiness during the previous 10 minutes. The scale ranges from 1, which indicates "extremely alert", to 9, which indicates "extremely sleepy, can't stay awake". Higher numbers indicating sleepier and lower numbers more alert. In this outcome measure, data for participants who received placebo matched to "1 mg, 2.5 mg, 5 mg E2006" and matched to "10 mg, 25 mg, 50 mg, 100 mg, and 200 mg E2006", has been presented separately.
Time Frame: Day 1 (Pre-dose), Day 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: Placebo: Matched to 1, 2.5, 5 mg E2006 | Part A: Placebo: Matched to 10, 25, 50, 100, 200 mg E2006 | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 6 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
score on a scale
  Day 1 (Pre-dose) | 5.2 (1.83) | 2.8 (1.48) | 3.2 (0.98) | 3.8 (2.04) | 3.5 (2.88) | 3.0 (1.10) | 2.0 (1.10) | 2.3 (2.07) | 2.2 (0.98) | 2.5 (1.52)
  Maximum Change From Day 1 (Pre-dose) at Day 6: number analyzed (Participants) | 6 | 10 | 5 | 6 | 5 | 6 | 6 | 5 | 6 | 6
  Maximum Change From Day 1 (Pre-dose) at Day 6 | -0.8 (4.02) | 0.5 (2.95) | 0.0 (2.55) | -0.2 (3.13) | 0.8 (4.60) | 5.3 (1.21) | 4.8 (2.99) | 5.4 (3.44) | 6.0 (1.26) | 6.3 (1.86)

35. Secondary Outcome: Part A: Change From Day 1 in Waketime Questionnaire Parameters: How Long Did You Sleep Last Night at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm a lack of sleep disturbance. In this outcome measure, data for question "How long did you sleep last night" has been reported.
Time Frame: Day 1, Day 6
Population: PD analysis set included all participants who had sufficient PD data to derive at least one PD parameter. Here "number analyzed" signifies participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
minutes
  Day 1 | 457.7 (24.81) | 475.0 (12.25) | 443.3 (42.39) | 436.7 (36.29) | 473.3 (7.53) | 469.2 (26.54) | 438.3 (21.37) | 455.0 (48.06) | 434.2 (45.21)
  Change From Day 1 at Day 6: number analyzed (Participants) | 9 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Change From Day 1 at Day 6 | 3.0 (29.58) |  |  |  | -85.8 (82.12) | 10.8 (26.54) | 22.5 (32.52) | -4.2 (21.54) | -11.0 (79.23)

36. Secondary Outcome: Part A: Change From Day 1 in Waketime Questionnaire Parameters: Time to Fall Asleep Last Night at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm a lack of sleep disturbance. In this outcome measure, data for question "Time to fall asleep last night" has been reported.
Time Frame: Day 1, Day 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
minutes
  Day 1 | 13.2 (6.99) | 15.7 (9.73) | 17.2 (9.91) | 14.5 (10.17) | 15.0 (8.94) | 16.7 (7.53) | 15.8 (3.76) | 10.0 (5.48) | 15.0 (7.07)
  Change From Day 1 at Day 6: number analyzed (Participants) | 9 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Change From Day 1 at Day 6 | 2.1 (10.46) |  |  |  | 20.0 (39.37) | -4.7 (6.68) | -3.8 (5.49) | 4.2 (3.76) | 7.0 (27.93)

37. Secondary Outcome: Part A: Change From Day 1 in Waketime Questionnaire Parameters: Number of Awakening After Falling Asleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm a lack of sleep disturbance. In this outcome measure, data for question "Number of awakening after falling asleep" has been reported.
Time Frame: Day 1, Day 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
number of awakenings
  Day 1 | 1.1 (0.77) | 1.8 (0.75) | 1.3 (1.03) | 0.8 (0.75) | 0.5 (0.84) | 1.2 (0.98) | 0.8 (0.98) | 1.8 (0.41) | 1.8 (1.72)
  Change From Day 1 at Day 6: number analyzed (Participants) | 9 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Change From Day 1 at Day 6 | -0.6 (1.24) |  |  |  | 1.7 (1.97) | 0.3 (1.51) | 0.2 (0.41) | -0.7 (1.03) | -1.0 (1.79)

38. Secondary Outcome: Part A: Change From Day 1 in Waketime Questionnaire Parameters: Time Spent Awake After Falling Asleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm a lack of sleep disturbance. In this outcome measure, data for question "Time spent awake after falling asleep" has been reported.
Time Frame: Day 1, Day 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
minutes
  Day 1 | 4.6 (4.86) | 6.2 (3.76) | 16.8 (22.14) | 5.3 (7.53) | 1.7 (2.58) | 5.0 (4.47) | 5.0 (6.32) | 11.2 (5.60) | 6.7 (4.08)
  Change From Day 1 at Day 6: number analyzed (Participants) | 9 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Change From Day 1 at Day 6 | -1.9 (8.18) |  |  |  | 53.3 (53.82) | 5.0 (8.37) | 5.0 (4.65) | -3.0 (7.75) | -2.5 (4.37)

39. Secondary Outcome: Part A: Change From Day 1 in Waketime Questionnaire Parameters: Rate Quality of Your Sleep at Day 6
Description: Participants were asked to answer the following question using Waketime Questionnaire: How long did you sleep last night, number of awakening after falling asleep, time to fall asleep last night, time spent awake after falling asleep, rate quality of your sleep (using Likert scale, ranged from 0 = very sound or restful, to 4 = very restless where lower score indicates better outcome). The primary purpose of the Waketime Questionnaire was to confirm a lack of sleep disturbance. In this outcome measure, data for question "Rate quality of your sleep" has been reported.
Time Frame: Day 1, Day 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
score on a scale
  Day 1 | 1.1 (0.77) | 0.3 (0.52) | 1.5 (1.22) | 0.7 (0.82) | 1.0 (0.00) | 0.5 (0.84) | 1.0 (0.89) | 0.8 (0.98) | 1.5 (0.84)
  Change From Day 1 at Day 6: number analyzed (Participants) | 9 | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6
  Change From Day 1 at Day 6 | 0.2 (0.67) |  |  |  | 1.3 (1.03) | 0.0 (0.00) | 0.0 (0.00) | 0.2 (0.75) | -0.2 (1.17)

40. Secondary Outcome: Part B: Number of Participants With Treatment Emergent Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs)
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
Participants
  AEs | 1 | 6 | 2 | 6 | 6
  SAEs | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Part B: Number of Participants With Markedly Abnormal Laboratory Parameter Values
Time Frame: Baseline up to Day 6
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
Participants | 3 | 6 | 4 | 3 | 7

42. Secondary Outcome: Part B: Number of Participants With Significant Change From Baseline in Vital Sign Values
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
Participants | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Part B: Number of Participants With Clinically Significant Change From Baseline in ECG Parameter Values
Time Frame: Baseline up to Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
Participants | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Part B: Number of Participants With Any Suicidality Assessed Using Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment [C-CASA]) is an interview-based rating scale to systematically assess any suicidality, any suicidal Behavior, any suicidal ideation. Any suicidality: emergence of any suicidal ideation or suicidal behavior. Any suicidal behavior: when response is "yes" for any these questions- actual attempt to suicide, engaged in non-suicidal self-injurious, behavior, interrupted attempt, aborted attempt, preparatory acts. Any suicidal ideation: when response is "yes" for any of these questions-wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent to suicide. Number of participants with any suicidality has been reported for this outcome measure.
Time Frame: Baseline, Day 11
Population: Safety analysis set included all participants who received study drug and had at least one postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
Number analyzed (Participants) | 12 | 11 | 13 | 10 | 12
Participants
  Baseline | 2 | 0 | 0 | 0 | 0
  Day 11 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 11 (for Both Part A and Part B)
Arm/Group | Part A: E2006 Matched Placebo | Part A: E2006 1.0 mg | Part A: E2006 2.5 mg | Part A: E2006 5 mg | Part A: E2006 10 mg | Part A: E2006 25 mg | Part A: E2006 50 mg | Part A: E2006 100 mg | Part A: E2006 200 mg | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo | Part B: Zolpidem 10 mg | Part B: E2006 2.5 mg | Part B: E2006 10 mg | Part B: E2006 25 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/11 | 0/13 | 0/10 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/11 | 0/13 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 7/16 | 1/6 | 0/6 | 1/6 | 4/6 | 2/6 | 4/6 | 2/6 | 5/6 | 1/12 | 6/11 | 2/13 | 6/10 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: E2006 Matched Placebo (N=16) | Part A: E2006 1.0 mg (N=6) | Part A: E2006 2.5 mg (N=6) | Part A: E2006 5 mg (N=6) | Part A: E2006 10 mg (N=6) | Part A: E2006 25 mg (N=6) | Part A: E2006 50 mg (N=6) | Part A: E2006 100 mg (N=6) | Part A: E2006 200 mg (N=6) | Part B: E2006 Matched Placebo or Zolpidem Matched Placebo (N=12) | Part B: Zolpidem 10 mg (N=11) | Part B: E2006 2.5 mg (N=13) | Part B: E2006 10 mg (N=10) | Part B: E2006 25 mg (N=12)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Application site erythema (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site irritation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Application site erosion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Euphoric mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypnagogic hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other